CLINICAL TRIAL: NCT06852950
Title: Continuous Glucose Monitoring for Outpatient Diabetes Management After Hospital Discharge
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Angel Morvant, Principal Investigator, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 242071
Record Dates: First submitted 2025-02-20; First posted 2025-02-28 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Type 2 Diabetes Mellitus (T2DM); Type 1 Diabetes Mellitus (T1DM); Hyperglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1; Hyperglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Libre 3 Plus Continuous Glucose Monitor (Experimental): Subjects in this arm will start using the Libre 3 Plus continuous glucose monitor.
  Interventions: Device: Libre 3 Plus Continuous Glucose Monitor
- Dexcom G7 Continuous Glucose Monitor (Experimental): Subjects in this arm will start using the Dexcom G7 continuous glucose monitor.
  Interventions: Device: Dexcom G7 Continuous Glucose Monitor

INTERVENTIONS:
Device: Libre 3 Plus Continuous Glucose Monitor — Subjects in this arm will start using the Libre 3 Plus continuous glucose monitor.
  Arms: Libre 3 Plus Continuous Glucose Monitor
Device: Dexcom G7 Continuous Glucose Monitor — Subjects in this arm will start using the Dexcom G7 continuous glucose monitor.
  Arms: Dexcom G7 Continuous Glucose Monitor

SUMMARY:
This study aims to improve patient awareness of the utility of continuous glucose monitoring systems in blood glucose monitoring and to improve patient satisfaction regarding diabetes care, particularly in the matter of blood glucose monitoring, at the transitions of care from the inpatient setting to the ambulatory setting.

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant adults, ages greater than or equal to 18 years, admitted to VUMC
* Able to give informed consent
* Hyperglycemia requiring insulin therapy including subcutaneous insulin injection or continuous subcutaneous insulin infusion (patient's own insulin pump) during hospitalization and at the time of discharge
* POC glucose or venous glucose levels in the 24 hours prior to participation need to be 70-350 mg/dL
* Need glucose readings greater than or equal to one time per day
* Mental status and dexterity adequate to use Libre 3 Plus or Dexcom G7 sensors with Libre 3 or Dexcom G7 application on patient's smartphone

Exclusion Criteria:

* Currently using Libre 3 Plus or Dexcom G7 CGMS during hospitalization or have used Libre 3 Plus or Dexcom G7 CGMS in the past 3 months
* Does not have smartphone compatible with Libre 3 App or Dexcom G7 App
* Received chemotherapy during current hospitalization
* Planning on major surgery within 10-15 days
* Hemodialysis or peritoneal dialysis
* Requiring vasopressors, intubation, sedation, or admission to an intensive care unit
* Vitamin C use of more than 500 milligrams per day
* Hydroxyurea use
* Acetaminophen use of more than 4 grams per day or 1 gram every 6 hours
* Significant pitting edema (3+ or greater) i.e. cirrhosis with ascites, congestive heart failure with edema, nephrotic syndrome, or signs of poor perfusion
* Presentation in diabetic ketoacidosis or hyperosmotic nonketotic state
* Skin allergy to adhesives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-09 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Questionnaire responses regarding patient satisfaction and opinion regarding use of continuous glucose monitoring system | From enrollment until follow-up telephone visit 2-3 weeks after discharge
  Questionnaire responses regarding patient satisfaction and opinion regarding use of continuous glucose monitoring system: regarding how do subjects feel that using CGM impacted their glucose control on a scale of 1-5, with 1=strongly made it worse, 2=somewhat made it worse, 3=did not make it better or worse, 4=somewhat made it better, and 5=strongly made it better?; regarding what is the overall opinion of subject's experience with CGM use on a scale of 1-5, with 1=very negative, 2=negative, 3=neutral, 4=positive, 5=very positive.
Questionnaire responses regarding patient satisfaction and opinion regarding quality of diabetes care | From enrollment until follow-up telephone visit 2-3 weeks after discharge
  Questionnaire responses regarding patient satisfaction and opinion regarding quality of diabetes care: regarding how do subjects feel that using CGM impacted the diabetes care overall on a scale of 1-5, with 1=strongly made it worse, 2=somewhat made it worse, 3=did not make it better or worse, 4=somewhat made it better, and 5=strongly made it better.
Questionnaire responses regarding patient familiarity with continuous glucose monitoring | From enrollment until follow-up telephone visit 2-3 weeks after discharge
  Questionnaire responses regarding patient familiarity with continuous glucose monitoring: regarding degree of familiarity of CGMs in general and the different types of information provided by CGMs, what is the subject's familiarity on a scale of 1-5, with 1=very unfamiliar, 2=unfamiliar, 3=neutral, 4=familiar, 5=very familiar.

SECONDARY OUTCOMES:
Degree of Average Change in Hemoglobin A1C from Start to End of Study | From enrollment until follow-up telephone visit 2-3 weeks after discharge
  Degree of average change in Hemoglobin A1C from start to end of study
Degree of Average Change in Glucose Management Indicator (GMI) | From enrollment until follow-up telephone visit 2-3 weeks after discharge
  Degree of average change in glucose management indicator (GMI)
Number of Participants with 30-day Readmissions Related to Glycemic Control | From enrollment until follow-up telephone visit 2-3 weeks after discharge
  Number of participants with 30-day Readmissions Related to Glycemic Control (hyperglycemia, hypoglycemia, or diabetic ketoacidosis)

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No